CLINICAL TRIAL: NCT02514291
Title: Evaluation of a Clinic-based Sleep Intervention for Pediatric Epilepsy
Brief Title: Sleep Intervention for Pediatric Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201412211RINA
Record Dates: First submitted 2015-07-28; First posted 2015-08-03 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2017-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep intervention (Experimental): Standard pediatric neurology care plus education and augmented support around adequate sleep habits, appropriate daylight exposure, and beneficial and safe physical activity tailored to each epileptic child's capabilities.
  Interventions: Behavioral: Sleep intervention
- Standard care (No Intervention): Standard pediatric neurology care

INTERVENTIONS:
Behavioral: Sleep intervention — Standard pediatric neurology care plus education and augmented support around adequate sleep habits, appropriate daylight exposure, and beneficial and safe physical activity tailored to each epileptic child's capabilities.
  Arms: Sleep intervention

SUMMARY:
The purpose of the study is to develop and evaluate a sleep intervention program for improving sleep and health in youth with epilepsy and their parents.

DETAILED DESCRIPTION:
Sleep problems are more prevalent and serious in children with epilepsy whose sleep can be disrupted by seizures occurring during the night and/or during the day. Inadequate sleep has long been recognized as a trigger for seizure and poor sleep habits have been associated with unfavorable outcomes in children with epilepsy. Attention to sleep in children with epilepsy as a result is critically important for seizure control and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1.5 and 6 years with a confirmed diagnosis of epilepsy based on clinical and electro-encephalogram examinations.

Exclusion Criteria:

* Children born before 37 weeks gestation, children with evidence of structural brain damage, or with cerebral palsy or those who are bedridden.

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Objective sleep | 12-month follow-up
  Actigraphic assessed sleep variables

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Tsai, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsai SY, Lee WT, Lee CC, Jeng SF, Weng WC. Behavioral-educational sleep interventions for pediatric epilepsy: a randomized controlled trial. Sleep. 2020 Jan 13;43(1):zsz211. doi: 10.1093/sleep/zsz211. PMID 31552428
- [Derived] Tsai SY, Lee WT, Lee CC, Jeng SF, Weng WC. Sleep in children with epilepsy: the role of maternal knowledge of childhood sleep. Sleep. 2018 Nov 1;41(11). doi: 10.1093/sleep/zsy157. PMID 30137598